CLINICAL TRIAL: NCT03472131
Title: Unilateral Posterolateral Approach for Disc Debridement and Titanium Cage Insertion Supplemented by Contralateral Transfascial Screw Fixation for Sick Patients Suffering From Septic Thoracolumbosacral Spondylodiscitis
Brief Title: Unilateral Posterolateral Approach for Spondylodiskitis
Acronym: SPDTIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Collaborators: St. Andrew's General Hospital, Patras, Greece (Other)
Responsible Party: Principal Investigator, Vasileios Syrimpeis, Orthopaedic Surgeon, University Hospital of Patras
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPONDYLODISKITIS2018
Record Dates: First submitted 2018-03-04; First posted 2018-03-21 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Discitis
Keywords: Spondylodiscitis; Titanium Cage; Posterolateral Debridement; Immunosuppressed; Less Invasive; Spine Infection
MeSH Terms: conditions — Discitis | interventions — Debridement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Septic spondylodiscitis (Experimental): A unilateral posterolateral approach and debridement with titanium cage insertion supplemented by screw fixation for severe sick patients suffering from septic spondylodiscitis
  Interventions: Procedure: Unilateral Posterolateral Approach and Debridement; Other: Titanium cage insertion supplemented by screw fixation

INTERVENTIONS:
Procedure: Unilateral Posterolateral Approach and Debridement
Other: Titanium cage insertion supplemented by screw fixation

SUMMARY:
This retrospective study assess the efficacy and safety of a posterolateral unilateral approach for debridement and titanium cage insertion supplemented by contralateral transfascial screw fixation for sick patients suffering from septic thoracolumbosacral spondylodiskitis. Hematogenous pyogenic spondylodiskitis requires surgical intervention in cases of development of neurological signs, spinal instability, progressive spinal deformity and abscess. When operative treatment is indicated, an anterior approach by open thoracotomy or by a thoraco-abdominal approach or combined anterior and posterior approaches are recommended. In cases of severe sick patients anterior approach is associated with high morbidity and mortality.

DETAILED DESCRIPTION:
Twenty consecutive sick (ASA>III) patients, 14 men and 6 women, aged 64±14 years, suffering from single level septic thoracolumbosacral spondylodiskitis underwent an one-stage less invasively unilateral posterolateral decompression, insertion of titanium cage& pedicle screw fixation plus contralateral transfascial pedicle screw fixation.

ELIGIBILITY:
Inclusion Criteria:

* Single-level thoracic, thoracolumbar, lumbar or lumbosacral spondylodiskitis
* Medical comorbidities were present in all 20 patients. These included diabetes mellitus, chronic renal insufficiency, advanced heart insufficiency, hypertension, cortisone abuse, drug abuse and/or advanced age (>65y).

Exclusion Criteria:

-

Ages: 44 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The extent of spinal cord injury (SCI) defined by the American Spinal Injury Association (ASIA) Impairment Scale | 2 years
  Grade A Complete lack of motor and sensory function below the level of injury (including the anal area) Grade B Some sensation below the level of the injury (including anal sensation) Grade C Some muscle movement is spared below the level of injury, but 50 percent of the muscles below the level of injury cannot move against gravity.
  Grade D Most (more than 50 percent) of the muscles that are spared below the level of injury are strong enough to move against gravity.
  Grade E All neurologic function has returned.

SECONDARY OUTCOMES:
Survival rate at 2,5 years | 2,5 years
  Revision surgery or "worst case scenario"
Survival rate at 10 years | 10 years
  Revision surgery or "worst case scenario"

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Korovessis, PhD, Principal Investigator — General Hospital of Patras

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Korovessis P, Syrimpeis V, Tsekouras V, Baikousis A, Vardakastanis K, Fennema P. A unilateral less invasive posterolateral approach for disc debridement and titanium cage insertion supplemented by contralateral transfascial screw fixation for high-morbidity patients suffering from septic thoracolumbosacral spondylodiscitis. Eur J Orthop Surg Traumatol. 2019 Aug;29(6):1187-1197. doi: 10.1007/s00590-019-02434-2. Epub 2019 Apr 16. PMID 30993521